CLINICAL TRIAL: NCT02540876
Title: A Pilot Study for Ilorasertib (ABT-348) in Patients With CDKN2A-deficient Advanced Solid Cancers: A Series of Individual Patient Cross-Over Studies With Growth Trajectory Assessment
Brief Title: Ilorasertib in Treating Patients With CDKN2A-deficient Advanced or Metastatic Solid Cancers That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-0083; NCI-2015-01328 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AbbVie IIS-10750; IRB15-0083 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Malignant Neoplasm; Solid Neoplasm; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ilorasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ilorasertib) (Experimental): Patients receive ilorasertib PO BID on days 1, 8, 15, 29, and 36. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ilorasertib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ilorasertib — Given PO
  Other Names: A-968660.0; ABT-348
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase I trial studies how well ilorasertib works in treating patients with cyclin-dependent kinase inhibitor 2A (CDKN2A)-deficient solid cancers that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or have spread to other places in the body (metastatic) and cannot be removed by surgery. Ilorasertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and consent to the Institutional Review Board (IRB) 13-0002 registry trial protocol
* Subjects must have histologically confirmed solid malignancy that is metastatic or unresectable
* The patient should have received all established therapies where there is a clear, superior available regimen available for the patient and the patient should have demonstrated progressive disease on or since completion of the last treatment regimen
* Patients must have measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral CT scan
* Patients must have prior CT scan images available for investigators to collect
* Patients must have available tumor molecular profiling from Clinical Laboratory Improvement Amendments (CLIA)-certified labs or have available archived tissue to be sent to such a laboratory in the context of this investigation
* Molecular testing in a CLIA-certified laboratory must have demonstrated a deletion involving the CDKN2A locus or a mutation within the locus that can be deemed from best available evidence to be likely to cause inactivation of a gene within or protein encoded by CDKN2A; sequencing or fluorescence in situ hybridization (FISH)/chromogenic in situ hybridization (CISH) methods are acceptable; the investigators will consider analyses performed according to similar standards as applied by Foundation Medicine (likely to be the most common source of molecular diagnostic data for patients in this trial)
* At least 3 weeks must have passed since any prior anti-tumor therapies including chemotherapy, radiation therapy or any other anti-cancer treatments
* Serum creatinine value of < 1.5 times the upper limit of normal (ULN) and either an estimated creatinine clearance value of > 50 mL/min as determined by the Chronic Kidney Disease Epidemiology (CKD EPI) or MDRD (Modification of Diet in Renal Disease) formulae or a creatinine clearance value of > 50 mL/min based on a 24 hour urine collection
* Subject has adequate liver function as demonstrated by serum bilirubin < 2 x ULN and Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN. For subjects with liver metastasis, adequate liver function is demonstrated by serum bilirubin =< 2 x ULN and AST/ALT =< 5.0 x ULN
* Subject has adequate bone marrow as demonstrated by absolute neutrophil count (ANC) >= 1,500/mm^3 (1.5 x 10^9/L); platelets >= 100,000/mm^2 (100 x 10^9/L); hemoglobin >= 9.0 g/dL (1.4 mmol/L)
* Subject has QTc interval < 500 msec on baseline electrocardiogram
* Subject has blood pressure controlled to < 150 mmHg systolic and < 95 mmHg diastolic at screening
* Subject has a documented left ventricular ejection fraction > 50%
* Women of child-bearing potential and men must agree to use adequate contraception (one of the following listed below) prior to the study entry, for the duration of study participation and up to 3 months following completion of therapy; women of child-bearing potential must have a negative pregnancy test within 7 days prior to initiation of treatment and post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential

  * Acceptable contraception

    * Total abstinence from sexual intercourse (minimum one complete menstrual cycle)
    * Vasectomized male subjects or vasectomized partner of female subjects
    * Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
    * Additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 3 months following completion of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-1
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients with hospitalization within 4 weeks of treatment initiation date for co-morbid conditions or any complication of disease or therapy that is deemed by the principal investigator as unstable or incompletely treated
* Patients with any psychiatric or social condition that leads them to be unlikely to adhere to the study schedule and contribute to the primary objectives
* Women that are pregnant or lactating are excluded from this study
* Subject has known active central nervous system (CNS) involvement; the subject has untreated brain or meningeal metastases; CT scans are not required to rule out brain or meningeal metastases unless there is a clinical suspicion of central nervous system disease; subjects with treated brain metastases that are radiographically or clinically stable for at least 4 weeks after therapy and have no evidence of cavitation or hemorrhage in the brain lesion(s) are eligible, providing that they are asymptomatic, and do not require corticosteroids (must have discontinued steroids at least 1 week prior to study drug administration)
* Subject has had major surgery within 28 days prior to study day 1
* Subject has proteinuria defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version [v] 4.0) grade > 1 at baseline as measured by a urine dipstick (2+ or greater) and confirmed by a 24 hour urine collection (>= 1 g/24 hrs); subjects may be re-screened if proteinuria is shown to be controlled with or without intervention
* Subject is taking any oral anticoagulant
* History of:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia (subjects with stable atrial fibrillation are not excluded)
  * Adrenal insufficiency
* Subject is unable to swallow or absorb oral tablets normally
* Subject takes cytochrome P450, family 3, subfamily A (CYP3A) inhibitors within 3 days or inducers within 7 days prior to the study drug administration; any questions or clarifications of these determinations should be brought to the attention of the principal investigator (PI); the PI will make the final determination on when it is safe to initiate ABT-348 (ilorasertib) therapy under circumstances where the magnitude or relevance of possible CYP3A4 inhibitors/inducers is unclear in the protocol appendix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Change in tumor burden. | 22 weeks
  Change in tumor measurements from baselines through end of study.

SECONDARY OUTCOMES:
Number of patients with response as per Response Evaluation Criteria in Solid Tumors (RECIST). | Up to week 12
  The number of patients with RECIST response will be estimated at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sharma, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States